CLINICAL TRIAL: NCT06876727
Title: A Target Trial Emulation for Efficacy and Safety of Antiplatelet Therapy After Endovascular Aortic Repair
Brief Title: Efficacy and Safety of Antiplatelet Therapy After Endovascular Aortic Repair
Acronym: EVAR_DAPT_SAPT
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: Antiplatelet After EVAR
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysms (AAA); Endovascular Aneurysm Repair (EVAR)
Keywords: Abdominal Aortic Aneurysms (AAA); Endovascular Aneurysm Repair (EVAR); Single antiplatelet therapy; Dual antiplatelet therapy
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dual antiplatelet therapy: Patients who were prescribed dual antiplatelet therapy at the date of discharge from the index hospitalization for standard EVAR
- Single antiplatelet therapy: Patients who were prescribed single antiplatelet therapy at the date of discharge from the index hospitalization for standard EVAR

SUMMARY:
This study was a target trial emulation using the National Health Claims database established by the Korean National Health Insurance Service (K-NHIS). 8,325 patients were included.

DETAILED DESCRIPTION:
Among these patients, any patients who were prescribed SAPT or DAPT at the date of discharge from the index hospitalization for standard EVAR were defined as being in the SAPT group (N=4,162) and the DAPT group (N=4,163), respectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent EVAR for AAA and were successfully discharged

Exclusion Criteria:

* Patients who had experienced a myocardial infarction
* Patients who had experienced a stroke
* Patients who had experienced percutaneous coronary intervention
* Patients who had history of peripheral disease
* Patients who had major bleeding event within 1 year of admission
* Those prescribed non-vitamin K antagonist oral anticoagulant or warfarin
* Patients who did not prescribe any antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent EVAR for AAA and were successfully discharged and prescribe any antiplatelet therapy.
Sampling Method: Non-Probability Sample
Enrollment: 8325 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 1 year after EVAR
  composite of all-cause death, myocardial infarction (MI), or ischemic stroke
Major or clinically relevant non-major bleeding | 1 year after EVAR
  Diagnostic codes in the primary or secondary position and transfusion receipt
Re-intervention or surgery for AAAs | 1 year after EVAR
  Re-intervention or surgery for AAAs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi KH, Kang D, Nam J, Park TK, Song MG, Seo TS, Yang WJ, Choi SH. Efficacy and Safety of Antiplatelet Therapy After Endovascular Aortic Repair: A Target Trial Emulation. J Am Heart Assoc. 2025 Oct 21;14(20):e044102. doi: 10.1161/JAHA.125.044102. Epub 2025 Oct 9. PMID 41065286